CLINICAL TRIAL: NCT00147030
Title: Whole Body Hypothermia for the Treatment of Perinatal Asphyxial Encephalopathy
Brief Title: TOBY (TOtal Body hYpothermia): a Study of Treatment for Perinatal Asphyxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISRCTN89547571(1)
Record Dates: First submitted 2005-09-05; First posted 2005-09-07 (Estimated); Results first posted 2016-05-11 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2013-11

CONDITIONS: Asphyxia Neonatorum; Hypoxia; Encephalopathy; Seizures
Keywords: Hypoxia; Ischaemia; Encephalopathy; Neonatal; Hypothermia; Perinatal; Cooling; Whole/Total Body
MeSH Terms: conditions — Asphyxia Neonatorum; Hypoxia; Brain Diseases; Seizures; Ischemia; Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cooled (Active Comparator): Whole body mild induced hypothermia for 72 hours, starting by 6 hours of age, in addition to standard intensive care. After 72 hours of cooling, rewarming by a maximum of 0.5 degree C / hour to normothermia.
  Interventions: Procedure: Whole body mild induced hypothermia
- non-cooled (No Intervention): Standard intensive care

INTERVENTIONS:
Procedure: Whole body mild induced hypothermia — Target rectal temperature 33-34°C for 72 hours, commencing by 6 hours of age; followed by re-warming at 0.5°C to normothermia
  Arms: cooled

SUMMARY:
Hypothesis: Prolonged whole body cooling in term infants with perinatal asphyxial encephalopathy reduces death and severe neurodevelopmental disability.

This study aims to determine whether whole body cooling to 33-34°C is a safe treatment that improves survival, without severe neurological or neurodevelopmental impairments at 18 months, of term infants suffering perinatal asphyxial encephalopathy.

DETAILED DESCRIPTION:
This is a multicentre prospective randomised controlled trial to determine whether a reduction of body temperature by 3-4°C following perinatal asphyxia improves survival without neurodevelopmental disability.

Full term infants will be randomised within 6 hours of birth to either a control group with the rectal temperature kept at 37 ± 0.2°C or to whole body cooling with the rectal temperature kept at 33.5 ± 0.5°C for 72 hours followed by slow rewarming.

The outcome will be assessed at 18 months of age by survival and neurological and neurodevelopmental testing.

Eligibility criteria:

Term infants less than 6 hours after birth with moderate or severe perinatal asphyxia (a combination of clinical and EEG criteria).

Exclusion criteria:

Infants expected to be 6 hours of age at the time of randomisation or infants with major congenital abnormalities.

Intervention:

Intensive care with whole body cooling versus intensive care without whole body cooling (babies are cooled to 33.5°C for 72 hours)

Main Outcomes:

Death and severe neurodevelopmental impairment at 18 months of age

Secondary Outcomes:

Cerebral thrombosis or haemorrhage, persistent hypotension, pulmonary hypertension, abnormal coagulation, arrhythmia and sepsis in the neonatal period. Neurological impairments at 18 months

Number of patients required: 236.

On 30th November 2006, when recruitment closed, 325 babies had been recruited.

ELIGIBILITY:
Inclusion criteria

The infant will be assessed sequentially by criteria A, B and C listed below:

A. Infants =>36 completed weeks gestation admitted to the Neonatal Intensive Care Unit (NICU) with at least one of the following:

* Apgar score of =<5 at 10 minutes after birth
* Continued need for resuscitation, including endotracheal or mask ventilation, at 10 minutes after birth
* Acidosis within 60 minutes of birth (defined as any occurrence of umbilical cord, arterial or capillary pH <7.00)
* Base Deficit =>16 mmol/L in umbilical cord or any blood sample (arterial, venous or capillary) within 60 minutes of birth

Infants that meet criteria A will be assessed for whether they meet the neurological abnormality entry criteria (B) by trained personnel:

B. Moderate to severe encephalopathy, consisting of altered state of consciousness (lethargy, stupor or coma) AND at least one of the following:

* hypotonia
* abnormal reflexes including oculomotor or pupillary abnormalities
* absent or weak suck
* clinical seizures

Infants that meet criteria A & B will be assessed by amplitude-integrated electroencephalogram (aEEG) (read by trained personnel):

C. At least 30 minutes duration of amplitude integrated EEG recording that shows abnormal background aEEG activity or seizures. There must be one of the following:

* normal background with some seizure activity
* moderately abnormal activity
* suppressed activity
* continuous seizure activity

Exclusion criteria

* Infants expected to be > 6 hours of age at the time of randomisation
* Major congenital abnormalities, such as diaphragmatic hernia requiring ventilation, or congenital abnormalities suggestive of chromosomal anomaly or other syndromes that include brain dysgenesis

Ages: 1 Hour to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 325 (Actual)
Dates: Start 2002-12; Primary Completion 2006-11 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denis Azzopardi, MD; FRCPCH, Principal Investigator — Imperial College London
Locations (1):
- Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Azzopardi DV, Strohm B, Edwards AD, Dyet L, Halliday HL, Juszczak E, Kapellou O, Levene M, Marlow N, Porter E, Thoresen M, Whitelaw A, Brocklehurst P; TOBY Study Group. Moderate hypothermia to treat perinatal asphyxial encephalopathy. N Engl J Med. 2009 Oct 1;361(14):1349-58. doi: 10.1056/NEJMoa0900854. PMID 19797281
- [Result] Rutherford M, Ramenghi LA, Edwards AD, Brocklehurst P, Halliday H, Levene M, Strohm B, Thoresen M, Whitelaw A, Azzopardi D. Assessment of brain tissue injury after moderate hypothermia in neonates with hypoxic-ischaemic encephalopathy: a nested substudy of a randomised controlled trial. Lancet Neurol. 2010 Jan;9(1):39-45. doi: 10.1016/S1474-4422(09)70295-9. Epub 2009 Nov 5. PMID 19896902

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Infants who met trial entry criteria were recruited at 40 Neonatal Intensive Care Units mainly in the United Kingdom and also in Europe. Recruitment took place over 4 years, from December 2006 to November 2006.
Pre-assignment Details: 494 infants were assessed for eligibility; 94 did not meet inclusion criteria, 30 declined to participate 45 were not enrolled for other reasons. 325 underwent randomization.
Groups:
- Non-cooled: Standard intensive care at normothermia
Period: Overall Study
Arm/Group | Cooled | Non-cooled
Started | 163 | 162
Completed | 163 | 162
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Infants who were less than 6 hours of age who had a gestational age of at least 36 weeks and perinatal asphyxial encephalopathy confirmed by 30 minutes' amplitude-integrated electro-encephalography that showed abnormal background activity or seizures.
Groups:
- Cooled: Whole body mild induced hypothermia 72 hours, commencing by 6 hours of age followed by re-warming to normothermia.
- Total: Total of all reporting groups
Arm/Group | Cooled | Non-cooled | Total
Number analyzed (Participants) | 163 | 162 | 325
Age, Customized [Number; unit: participants] — All participants were < 6 hours of age at randomization.
  participants
    Age 0-4 hours | 48 | 57 | 105
    Age 4-6 hours | 115 | 105 | 220
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 74 | 136
  Male | 101 | 88 | 189

OUTCOME MEASURES:

1. Primary Outcome: Combined Incidence of Mortality and Severe Neurodevelopmental Disability in Survivors
Description: Severe neurodevelopmental disability was defined as a score of less than 70 on the Mental Developmental Index of the Bayley Scales of Infant Development II (BSID-II) (on which the standardization mean [± standard deviation (SD)] is 100±15 and higher scores indicate better performance), a score of 3 to 5 on the Gross Motor Function Classification System (GMFCS) (on which scores can range from 1 to 5, with higher scores indicating greater impairment), or bilateral cortical visual impairment with no useful vision.
Time Frame: 18 months
Measure: Number; unit: participants
Groups:
- Cooled: Whole body mild induced hypothermia commencing by 6 hours of age for 72 hours, followed by normothermia.
Arm/Group | Cooled | Non-cooled
Number analyzed (Participants) | 163 | 162
participants | 74 | 86

2. Secondary Outcome: Intracranial Haemorrhage
Description: Intracranial hemorrhage was identified on magnetic resonance imaging (MRI).
Time Frame: Duration of hospital stay, on average 22 days
Measure: Number; unit: participants
Groups:
- Cooled: Whole body mild induced hypothermia commencing by 6 hours of age for 72 hours; followed by normothermia.
Arm/Group | Cooled | Non-cooled
Number analyzed (Participants) | 64 | 67
participants | 25 | 21

3. Secondary Outcome: Persistent Hypotension
Description: Hypotension was defined as a mean blood pressure of 40 mm Hg or less and was persistent if causes of hypotension had been sought and appropriate treatment provided, without success.
Time Frame: Duration of hospital stay, on average 22 days
Measure: Number; unit: participants
Arm/Group | Cooled | Non-cooled
Number analyzed (Participants) | 163 | 162
participants | 126 | 134

4. Secondary Outcome: Pulmonary Haemorrhage
Time Frame: Duration of hospital stay, on average 22 days
Measure: Number; unit: participants
Arm/Group | Cooled | Non-cooled
Number analyzed (Participants) | 163 | 162
participants | 5 | 3

5. Secondary Outcome: Pulmonary Hypertension
Time Frame: Duration of hospital stay, on average 22 days
Measure: Number; unit: participants
Arm/Group | Cooled | Non-cooled
Number analyzed (Participants) | 163 | 162
participants | 16 | 9

6. Secondary Outcome: Prolonged Blood Coagulation Time
Time Frame: Duration of hospital stay, on average 22 days
Measure: Number; unit: participants
Arm/Group | Cooled | Non-cooled
Number analyzed (Participants) | 163 | 161
participants | 67 | 72

7. Secondary Outcome: Culture Proven Sepsis
Time Frame: Duration of hospital stay, on average 22 days
Measure: Number; unit: participants
Arm/Group | Cooled | Non-cooled
Number analyzed (Participants) | 163 | 162
participants | 20 | 20

8. Secondary Outcome: Necrotising Enterocolitis
Time Frame: Duration of hospital stay, on average 22 days
Measure: Number; unit: participants
Arm/Group | Cooled | Non-cooled
Number analyzed (Participants) | 163 | 162
participants | 1 | 0

9. Secondary Outcome: Cardiac Arrhythmia
Description: Arrhythmia identified on electrocardiogram (ECG), e.g. sinus bradycardia <80 beats per minute, ventricular arrhythmia.
Time Frame: Duration of hospital stay, on average 22 days
Measure: Number; unit: participants
Arm/Group | Cooled | Non-cooled
Number analyzed (Participants) | 163 | 162
participants | 8 | 3

10. Secondary Outcome: Thrombocytopenia
Time Frame: Duration of hospital stay, on average 22 days
Measure: Number; unit: participants
Arm/Group | Cooled | Non-cooled
Number analyzed (Participants) | 163 | 161
participants | 94 | 80

11. Secondary Outcome: Major Venous Thrombosis
Time Frame: Duration of hospital stay, on average 22 days
Measure: Number; unit: participants
Arm/Group | Cooled | Non-cooled
Number analyzed (Participants) | 163 | 162
participants | 2 | 1

12. Secondary Outcome: Renal Failure Treated With Dialysis
Time Frame: Duration of hospital stay, on average 22 days
Measure: Number; unit: participants
Arm/Group | Cooled | Non-cooled
Number analyzed (Participants) | 163 | 162
participants | 0 | 0

13. Secondary Outcome: Pneumonia
Time Frame: Before discharge from hospital
Measure: Number; unit: participants
Arm/Group | Cooled | Non-cooled
Number analyzed (Participants) | 163 | 162
participants | 5 | 5

14. Secondary Outcome: Pulmonary Airleak
Time Frame: Duration of hospital stay, on average 22 days
Measure: Number; unit: participants
Arm/Group | Cooled | Non-cooled
Number analyzed (Participants) | 163 | 162
participants | 9 | 3

15. Secondary Outcome: Duration of Hospitalisation
Description: Total duration of hospital care
Time Frame: Duration of hospital stay, on average 22 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Cooled | Non-cooled
Number analyzed (Participants) | 163 | 162
days | 12 [8 to 18] | 13 [9 to 25]

16. Secondary Outcome: Mortality
Time Frame: 18 months
Measure: Number; unit: participants
Arm/Group | Cooled | Non-cooled
Number analyzed (Participants) | 163 | 162
participants | 42 | 44

17. Secondary Outcome: Severe Neurodevelopmental Disability
Time Frame: 18 months
Population: Number of participants analyzed is reduced due to deaths prior to assessment and not all survivors could complete all elements of the examination. Number analyzed represents the participants on whom the relevant data for this outcome could be documented.
Measure: Number; unit: participants
Arm/Group | Cooled | Non-cooled
Number analyzed (Participants) | 120 | 117
participants | 32 | 42

18. Secondary Outcome: Multiple Handicap
Description: defined as the presence of any two of the following in an infant; neuromotor disability (Level 3-5 on Gross Motor Function classification), mental delay (Bayley Mental Developmental Index (MDI) score < 70), epilepsy, cortical visual impairment, sensorineural hearing loss
Time Frame: 18 months
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Cooled | Non-cooled
Number analyzed (Participants) | 112 | 110
participants | 21 | 33

19. Secondary Outcome: Bayley Psychomotor Developmental Index Score (PDI)
Description: Bayley Psychomotor Developmental Index score (PDI) <70
Time Frame: 18 months
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Cooled | Non-cooled
Number analyzed (Participants) | 114 | 109
participants | 27 | 37

20. Secondary Outcome: Sensorineural Hearing Loss
Description: Normal or near normal hearing, no sensorineural hearing loss
Time Frame: 18 months
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Cooled | Non-cooled
Number analyzed (Participants) | 120 | 117
participants | 110 | 97

21. Secondary Outcome: Epilepsy (Defined as Recurrent Seizures Beyond the Neonatal Period, Requiring Anticonvulsant Therapy at the Time of Assessment)
Time Frame: 18 months
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Cooled | Non-cooled
Number analyzed (Participants) | 116 | 116
participants | 12 | 16

22. Secondary Outcome: Microcephaly
Description: Head circumference at follow-up >2 standard deviations below the mean
Time Frame: 18 months
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Cooled | Non-cooled
Number analyzed (Participants) | 114 | 112
participants | 24 | 28

ADVERSE EVENTS:
Arm/Group | Cooled | Non-cooled
Serious Adverse Events (participants affected / at risk) | 8/163 | 3/162
Other Adverse Events (participants affected / at risk) | 126/163 | 134/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cooled (N=163) | Non-cooled (N=162)
Hypotension (Cardiac disorders) | 2 (2) | 2 (2) — Severe hypotension (mean arterial pressure less than 25mmHg), despite full inotrope support and volume replacement.
Cardia arrhythmia (Cardiac disorders) | 3 (3) | 2 (2)
Major venous thrombosis not related to an infusion line. (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Collapse (Surgical and medical procedures) | 1 (1) | 0 (0) — Collapse during lumbar puncture
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cooled (N=163) | Non-cooled (N=162)
Persistent hypotension (Cardiac disorders) | 126 | 134 — Hypotension was defined as a mean blood pressure of 40 mm Hg or less.
Prolonged coagulation time (Blood and lymphatic system disorders) | 67 | 72
Thrombocytopenia (Blood and lymphatic system disorders) | 94 | 80
Intracranial hemorrhage (Nervous system disorders) | 25 | 21
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Pulmonary air leak (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 16 | 9
Necrotizing enterocolitis (Gastrointestinal disorders) | 1 | 0
Culture-proven sepsis (Infections and infestations) | 20 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No